CLINICAL TRIAL: NCT03711487
Title: The Effect of Foeniculum Vulgare Ironing on Gastrointestinal Recovery After Colorectal Resection: a Randomized Controlled Trial.
Brief Title: The Effect of Foeniculum Vulgare Ironing on Gastrointestinal Recovery After Colorectal Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FV-GIR-2018
Record Dates: First submitted 2018-10-12; First posted 2018-10-18 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Surgery; Foeniculum; Ileus
Keywords: Colorectal surgery; Foeniculum; Ileus
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ironing therapy (Experimental): Stir-fry 500 grams of Foeniculum vulgare seeds until the aroma overflows. Put them into a cotton bag. Ironing therapy put the bag on abdomen after the temperature is suitable, 30 minutes per time, 4 times daily from 12 hours after surgery and last for 2 days. The medicine bag can be heated and reused after it cool down.
  Interventions: Drug: Foeniculum Vulgare Seed Ironing
- No intervention (No Intervention): No intervention.

INTERVENTIONS:
Drug: Foeniculum Vulgare Seed Ironing — Stir-fry 500 grams of Foeniculum vulgare seeds until the aroma overflows. Put them into a cotton bag. Ironing therapy put the bag on abdomen after the temperature is suitable, 30 minutes per time, twice daily on postoperative days 2 to 3. The medicine bag can be heated and reused after it cool down.
  Arms: Ironing therapy

SUMMARY:
Chinese Medicine Ironing using Foeniculum vulgare has been applied in some departments to promote bowel function recovery, but the efficacy of ironing therapy remains uncertain after colorectal resection surgery.

DETAILED DESCRIPTION:
Postoperative ileus is one of the most common complications after abdominal surgery. It refers to obstipation and intolerance of oral intake due to nonmechanical factors that disrupt the normal coordinated propulsive motor activity of the gastrointestinal tract following abdominal or nonabdominal surgery. When the expected period of gastrointestinal recovery time extends beyond what is acceptable, the patient is diagnosed as having a "pathologic" postoperative ileus (POI), which leads to patient discomfort, dissatisfaction, prolonged hospitalization and increased medical expenses. The incidence of POI is about 17%~24% after abdominal surgery. Chinese Medicine Ironing using Foeniculum vulgare has been applied in some departments to promote gastrointestinal function recovery as a empiric therapy. However, the definite efficacy of Foeniculum vulgare ironing therapy（FIT）is uncertain after colorectal resection surgery and whether FIT can reduce the incidence of POI remains unkonown.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 ~ 85 years old; sex is not limited.
2. Selective operation of colorectal partial resection.
3. Participants are volunteered to participate in this study, sign informed consent, and cooperated with follow-up.

Exclusion Criteria:

1. Emergency surgery.
2. Pregnant or lactating women.
3. ASA class 4 or 5 patients.
4. Patients with severe abdominal adhesions, which would cost more than 30 minutes to release. Patients with abdominal cocoon disease.
5. Patients with peritoneal metastasis or inflammatory bowel disease.
6. Patients undergoing enterostomy or total colectomy.
7. Patients simultaneously enrolled in any other competing clinical study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Flatus time | Up to 30 days after operation.
  Time to faltus (hours from end of operation). Patients who had stool before any movement of gas were deemed to have an equal time to the time to flatus and first bowel movement.
Incidence of postoperative ileus | 4 days after operation
  The same panel defined "prolonged" postoperative ileus as the occurrence of two or more of the following signs and symptoms on postoperative day 4 or after: Nausea or vomiting, Inability to tolerate an oral diet over the preceding 24 hours, Absence of flatus over the preceding 24 hours, Abdominal distention.

SECONDARY OUTCOMES:
Toleration of a low-residue diet | Up to 30 days after operation.
  Time (hours from end of operation) to tolerate a low-residue diet, defined as consuming >50% of the meal without emesis for 24 hours (time recorded was the time when the patient ate >50% of the meal).
Toleration of drinking water | Up to 30 days after operation.
  Time (hours from end of operation) to toleration of water.
Duration of postoperative hospitalization | Up to 30 days after operation.
  Postoperative days the patient was ready for hospital discharge based on Gastrointestinal function alone.
Pain assessment | During postoperative hospitalization, up to 30 days after operation.
  Assess postoperative pain with the pain visual analogue scale. Rate the pain levels on a likert scale from 0 (no pain) to 10 (pain as bad as it could possibly be).
Nausea and appetite assessment | During postoperative hospitalization, up to 30 days after operation.
  Rate their appetite and nausea levels on a likert scale from 0 (no appetite, nausea) to 10 (appetite as good as can be, nausea as bad as can be), and each score was recorded separately.
Short-term complications | Up to 30 days after operation.
  Complications during the 30-day postoperative period
Adverse events | Up to 30 days after operation.
  Any adverse events possibly related to treatment with Foeniculum vulgare ironing.
Hospitalization costs | During postoperative hospitalization, up to 30 days after operation.
  Postoperative in-patients costs

CONTACTS AND LOCATIONS:
Overall Officials: Ziqiang Wang, MD, Study Chair — West China Hospital
Locations (1):
- Guoxue Road 37#,West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choi EM, Hwang JK. Antiinflammatory, analgesic and antioxidant activities of the fruit of Foeniculum vulgare. Fitoterapia. 2004 Sep;75(6):557-65. doi: 10.1016/j.fitote.2004.05.005. PMID 15351109
- [Result] Iyer S, Saunders WB, Stemkowski S. Economic burden of postoperative ileus associated with colectomy in the United States. J Manag Care Pharm. 2009 Jul-Aug;15(6):485-94. doi: 10.18553/jmcp.2009.15.6.485. PMID 19610681
- [Result] Ma HW, Zhao JT, Zhao X. [The Effect of Fennel Tea Drinking on Postoperative Gut Recovery after Gynecological Malignancies Operation]. Sichuan Da Xue Xue Bao Yi Xue Ban. 2015 Nov;46(6):940-3. Chinese. PMID 26867333
- [Result] Miguel MG, Cruz C, Faleiro L, Simoes MT, Figueiredo AC, Barroso JG, Pedro LG. Foeniculum vulgare essential oils: chemical composition, antioxidant and antimicrobial activities. Nat Prod Commun. 2010 Feb;5(2):319-28. PMID 20334152
- [Result] Rezayat SM, Dehpour AR, Motamed SM, Yazdanparast M, Chamanara M, Sahebgharani M, Rashidian A. Foeniculum vulgare essential oil ameliorates acetic acid-induced colitis in rats through the inhibition of NF-kB pathway. Inflammopharmacology. 2018 Jun;26(3):851-859. doi: 10.1007/s10787-017-0409-1. Epub 2017 Oct 24. PMID 29067571
- [Result] Jang SH, Yang DK. The combination of Cassia obtusifolia L. and Foeniculum vulgare M. exhibits a laxative effect on loperamide-induced constipation of rats. PLoS One. 2018 Apr 5;13(4):e0195624. doi: 10.1371/journal.pone.0195624. eCollection 2018. PMID 29621360
- [Result] Mattei P, Rombeau JL. Review of the pathophysiology and management of postoperative ileus. World J Surg. 2006 Aug;30(8):1382-91. doi: 10.1007/s00268-005-0613-9. PMID 16850151
- [Result] Bragg D, El-Sharkawy AM, Psaltis E, Maxwell-Armstrong CA, Lobo DN. Postoperative ileus: Recent developments in pathophysiology and management. Clin Nutr. 2015 Jun;34(3):367-76. doi: 10.1016/j.clnu.2015.01.016. Epub 2015 Jan 31. PMID 25819420